CLINICAL TRIAL: NCT00966836
Title: Efficacy and Safety of Anti-cytomegalovirus Prophylaxis Versus Pre-emptive Approaches With Valganciclovir in Heart Transplant Recipients Treated With Everolimus or Mycophenolate. A Randomized Open-label Study for Prevention of Cardiaca Allograft Vasculopathy
Brief Title: Prevention of Transplant Atherosclerosis With Everolimus and Anti-cytomegalovirus Therapy
Acronym: PROTECT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Angelo Branzi, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROTECT 2008-006980-35
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: Heart Transplantation; Cardiac Allograft Vasculopathy; Cytomegalovirus Infection
Keywords: Heart Transplantation; Cardiac Allograft Vasculopathy; Cytomegalovirus Infection; Everolimus; Valganciclovir; Mycophenolate
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir; Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pre-emptive everolimus (Experimental)
  Interventions: Drug: Pre-emptive strategy with valganciclovir plus everolimus
- Prophylaxis mycophenolate (Experimental)
  Interventions: Drug: Prophylaxis with valganciclovir plus mycophenolate
- Prophylaxis Everolimus (Experimental)
  Interventions: Drug: Prophylaxis with valganciclovir plus everolimus
- Pre-emptive mycophenolate (Active Comparator)
  Interventions: Drug: Pre-emptive mycophenolate

INTERVENTIONS:
Drug: Pre-emptive strategy with valganciclovir plus everolimus — Patients will be monitored for CMV infection and receive valganciclovir only for positive PCR or antigenemia. Everolimus plus cyclosporine and prednisone will be used for maintenance immunosuppression
  Arms: Pre-emptive everolimus
Drug: Prophylaxis with valganciclovir plus mycophenolate — Patients will receive 3 months of oral valganciclovir with mycophenolate and standard cyclosporine and prednisone for maintenance immunosuppression
  Arms: Prophylaxis mycophenolate
Drug: Prophylaxis with valganciclovir plus everolimus — Patients will receive valganciclovir for 3 months after transplant. Everolimus plus reduced cyclosporine and prednisone will be used for maintenance immunosuppression
  Arms: Prophylaxis Everolimus
Drug: Pre-emptive mycophenolate — Patients will be monitored for CMV infection and receive valganciclovir only for positive PCR or antigenemia. Mycophenolate plus standard cyclosporine and prednisone will be used for maintenance immunosuppression
  Arms: Pre-emptive mycophenolate

SUMMARY:
Cardiac allograft vasculopathy (CAV) is the major cause of long-term graft failure in heart transplant recipients. Although several immune-mediated and metabolic risk factors have been implicated in the pathogenesis of CAV, no effective therapy is currently available to treat established CAV and prevent its adverse outcomes. Therefore, the main clinical strategy is based on prevention and treatment of factors known to trigger its development. Although the mechanism is vague, cytomegalovirus (CMV) infection is believed to play a key role in CAV progression.

Two strategies involving administration of specific anti-CMV agents are recommended for prevention of CMV infection/disease: universal prophylaxis and preemptive therapy. The pros and cons of the two strategies are still debated, in the absence of randomized studies addressing graft-related outcomes and viral mechanisms of graft damage, and without any clear evidence of superiority of either approach.

The investigators conceived this randomized prospective project to compare the effect of preemptive anti-CMV strategy with universal anti-CMV prophylaxis on CMV infection and on one-year increase in coronary intimal thickening. Patients will be additionally randomized to receive either mycophenolate mofetil or everolimus, in light of the possible anti-CMV properties of everolimus.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18y
* Heart or heart-kidney combined transplant
* Positive CMV serology at the time of transplant
* Glomerular filtration rate ≥ 20 ml/min/1.73m2 with MDRD at randomization.
* Written informed consent

Exclusion Criteria:

* Panel Reactive Antibody ≥50%
* Less than 1000/mmc neutrophils at the time of randomization
* Less than 30,000/mmc platelets at the time of randomization
* Clinical significant infection in the 2 weeks prior to transplant
* Glomerular filtration rate < 20 ml/min/1.73m2 estimated with MDRD formula at the time of randomization or hemodialysis treatment
* Intolerance towards valganciclovir, everolimus, mycophenolate or cyc-losporine
* Known contraindication to statin use
* Negative CMV serology at the time of transplant
* HIV positive testing
* Severe comorbidities that, based on investigator's judgment, contraindicate study drugs or procedures
* Potentially childbearing women who refuse to use contraceptives
* Participation to an interventional study in the 2 preceding weeks
* Unwillingness or inability to follow study procedure and to sign written in-formed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Change in maximal intimal thickness | one year

SECONDARY OUTCOMES:
CMV infection | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria S Orsola Malpighi, Bologna, Italy

REFERENCES:
- [Background] Potena L, Grigioni F, Magnani G, Lazzarotto T, Musuraca AC, Ortolani P, Coccolo F, Fallani F, Russo A, Branzi A. Prophylaxis versus preemptive anti-cytomegalovirus approach for prevention of allograft vasculopathy in heart transplant recipients. J Heart Lung Transplant. 2009 May;28(5):461-7. doi: 10.1016/j.healun.2009.02.009. PMID 19416774
- [Background] Potena L, Valantine HA. Cytomegalovirus-associated allograft rejection in heart transplant patients. Curr Opin Infect Dis. 2007 Aug;20(4):425-31. doi: 10.1097/QCO.0b013e328259c33b. PMID 17609604
- [Background] Hill JA, Hummel M, Starling RC, Kobashigawa JA, Perrone SV, Arizon JM, Simonsen S, Abeywickrama KH, Bara C. A lower incidence of cytomegalovirus infection in de novo heart transplant recipients randomized to everolimus. Transplantation. 2007 Dec 15;84(11):1436-42. doi: 10.1097/01.tp.0000290686.68910.bd. PMID 18091519
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045